CLINICAL TRIAL: NCT01379560
Title: A Study to Evaluate the Ocular Blood Flow Effects of Unoprostone Isopropyl in Adults With Dry Age-related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Sucampo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPA/UIOS-AMD-1021
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2013-03

CONDITIONS: Dry Age-related Macular Degeneration
MeSH Terms: interventions — isopropyl unoprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- unoprostone isopropyl (2 drop) (Experimental)
  Interventions: Drug: unoprostone isopropyl
- unoprostone isopropyl (3 drop) (Experimental)
  Interventions: Drug: unoprostone isopropyl

INTERVENTIONS:
Drug: unoprostone isopropyl — 1. unoprostone isopropyl (2 drops)
  2. placebo (2 drops)
  Arms: unoprostone isopropyl (2 drop)
Drug: unoprostone isopropyl — 1. unoprostone isopropyl (3 drops)
  2. placebo (3 drops)
  Arms: unoprostone isopropyl (3 drop)

SUMMARY:
The purpose of this study is to determine the pharmacodynamics of ocular blood flow measurements with multiple drop unoprostone isopropyl administration versus placebo in subjects with dry age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years at screening
* Ametropy ≤ 3 diopters
* Clear ocular media
* Visual acuity in the study eye > 20/40

Exclusion Criteria:

* Presence of any ocular condition in the study eye (other than AMD) that may progress during the course of the study and could affect central vision, or other ocular conditions that may be a confounding factor in this study
* Blood donation during the previous 3 weeks
* Current smoker or a history of smoking within 5 years of enrollment
* Treatment with protocol-specified prohibited concomitant medications
* Prior exposure to Rescula (unoprostone isopropyl) and or a known sensitivity to any of the components of the study medication (e.g. benzalkonium chloride)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in choroidal blood flow | In total 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria